CLINICAL TRIAL: NCT01310530
Title: Phase 2 Trial of Partial Breast Proton Therapy for Early Stage Breast Cancer With Low and Intermediate Risk Factors.
Brief Title: Partial Breast Proton Therapy for Early Stage Breast Cancer
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5110026
Record Dates: First submitted 2011-03-07; First posted 2011-03-08 (Estimated); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Partial Breast; Proton Beam
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Partial Breast Proton Therapy (Experimental): Two weeks of daily proton therapy delivered to the lumpectomy site.
  Interventions: Radiation: Proton Beam Radiotherapy

INTERVENTIONS:
Radiation: Proton Beam Radiotherapy — Daily proton beam radiotherapy is delivered to the site of the breast tumor in ten treatment sessions over two week as an outpatient.

SUMMARY:
The purpose of this is to determine the efficacy and toxicity of proton therapy when used to deliver partial breast radiotherapy in patients with early stage breast cancer with low or intermediate risk factors.

DETAILED DESCRIPTION:
Radiation therapy delivered to the whole breast is standard treatment following tumor removal for patients with early stage breast cancer. In selected patients, delivering the radiation treatment to only the part of the breast involved by the tumor may be a viable alternative. This can decrease the amount of normal tissues exposed to irradiation, potentially decrease side-effects and shorten the treatment time. Proton beam can decrease the volume of normal tissues treated compared to standard forms of radiotherapy. This study will recruit patients with early stage breast cancer following surgical removal to undergo partial breast radiotherapy with proton beam and determine the recurrence rates and side-effects of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Breast carcinoma
* DCIS
* Age 40 years or higher
* Primary tumor 3 cm or less
* Lumpectomy with clip placement
* Axillary node sampling
* Negative margins

Exclusion Criteria:

* Distant metastasis
* Multicentric disease
* Prior radiation or chemotherapy
* Active collagen vascular disease
* Pregnant or lactating
* BRCA mutation
* Lymph nodes with more than microscopic tumor involvement

Ages: 40 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-05-04 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Rate of recurrence in the breast | 5 years

SECONDARY OUTCOMES:
Rate of breast recurrence of low versus intermediate risk patients | 5 years
Side-effects related to treatment | 5 years
Disease Free Survival | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David A Bush, MD, Principal Investigator — Radiation Medicine - Loma Linda University Medical Center
Locations (2):
- United States (2):
  - Loma Linda University Medical Center / James M. Slater MD Proton Treatment Center / Department of Radiation Medicine / 11234 Anderson St., Loma Linda, California
  - Loma Linda University Medical Center, Loma Linda, California

REFERENCES:
- [Background] Bush DA, Slater JD, Garberoglio C, Yuh G, Hocko JM, Slater JM. A technique of partial breast irradiation utilizing proton beam radiotherapy: comparison with conformal x-ray therapy. Cancer J. 2007 Mar-Apr;13(2):114-8. doi: 10.1097/PPO.0b013e318046354b. PMID 17476139